CLINICAL TRIAL: NCT01191879
Title: A Comparison of p53-induced Genes Activation as Possible Markers Differentiating Between Patients Presenting With Acute Myocardial Infarction and Controls
Brief Title: A Comparison of p53-induced Genes Activation in Patients With and Without Acute Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MRNA-MI-1
Record Dates: First submitted 2010-08-08; First posted 2010-08-31 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Acute Myocardial Infarction
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- acute MI group: Patients presenting with acute ST elevation myocardial infarction, admitted to the intensive cardiac care unit and that are planned for emergency primary PCI
  Interventions: Other: Blood test
- Controls: Patients undergoing a non-invasive evaluation of possible myocardial ischemia.
  Interventions: Other: Blood test

INTERVENTIONS:
Other: Blood test — Blood test

SUMMARY:
The purpose of this study is to compare p53-induced genes activation as possible markers differentiating between patients presenting with acute myocardial infarction and controls.

DETAILED DESCRIPTION:
The diagnosis of acute myocardial infarction is based on the rise of bio-markers for cardiac necrosis such as troponin. While troponin measurement is highly sensitive for myocardial necrosis it has several limitations that influence its clinical use. First, since the troponin test is reliable only after 4-6 hours from symptoms onset, it has only limited value in the assessment of patients presenting earlier. Second, several clinical situations, most commonly renal dysfunction, are associated with increased troponin level and therefore may decrease the specificity of the test. Third, since troponin rise indicates myocardial infarction it is not useful in the common situations where there is myocardial ischemia without necrosis.

The P53 is a tumor suppressing gene activated in different stressful situations including hypoxia. This activation is associated with accelerated transcription (up to 30-50 folds from baseline) of different genes that are involved in apoptosis, DNA repair and in stopping the cell cycle. A study on pregnant women demonstrated high levels of fetal mRNA of these genes in maternal circulation. This gene expression correlated with other signs of fetal stress associated with hypoxia. Myocardial ischemia is another stressful event associated with tissue hypoxia. Nevertheless, the association of this gene expression with myocardial ischemia has not been investigated yet.

ELIGIBILITY:
Inclusion Criteria:

Acute MI group:

Patient presenting with chest pain lasting for at leasY 1 hour and no more than 6 hours accompanied by 1 of the following ECG criteria:

* ST segment elevation of anterior or inferior wall (at least 2 consecutive leads)
* New LBBB

Controls:

* Patients undergoing non-invasive evaluation of possible myocardial ischemia

Exclusion Criteria:

* Chronic lung disease requiring chronic treatment
* Any malignancy in the 5 year prior to enrollment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Aacute MI group- Patients with acute ST elevation MI planned for emergency primary PCI
  Controls: Patients undergoing non-invasive evaluation of possible myocardial ischemia
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2010-11; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Expression of P53 induced genes in patients with and without acute myocardial infarction | Up to 4 hours following recruitment

SECONDARY OUTCOMES:
Correlation between P53 associated gene expression with troponin level | After 5 days from recruitment

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel, Israel

REFERENCES:
- [Background] Ashur-Fabian O, Avivi A, Trakhtenbrot L, Adamsky K, Cohen M, Kajakaro G, Joel A, Amariglio N, Nevo E, Rechavi G. Evolution of p53 in hypoxia-stressed Spalax mimics human tumor mutation. Proc Natl Acad Sci U S A. 2004 Aug 17;101(33):12236-41. doi: 10.1073/pnas.0404998101. Epub 2004 Aug 9. PMID 15302922